CLINICAL TRIAL: NCT00005654
Title: Randomized Study of the Effect of Decreased Hyperinsulinemia on the Ovulatory Response to Clomiphene Citrate in Obese Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Virginia (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/14914; UVA-WSE023
Record Dates: First submitted 2000-05-02; First posted 2000-05-03 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-04

CONDITIONS: Hyperinsulinism; Polycystic Ovary Syndrome
Keywords: endocrine disorders; hyperinsulinism; polycystic ovarian syndrome; rare disease
MeSH Terms: conditions — Hyperinsulinism; Polycystic Ovary Syndrome; Endocrine System Diseases; Rare Diseases | interventions — Clomiphene; Metformin

INTERVENTIONS:
Drug: clomiphene citrate
Drug: metformin

SUMMARY:
OBJECTIVES:

I. Determine whether reduction of serum insulin levels by metformin increases ovulatory response to clomiphene or spontaneous ovulation in obese women with polycystic ovary syndrome.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are randomized to one of two treatment arms.

Patients receive oral metformin (arm I) or oral placebo (arm II) three times daily for 8 weeks. All patients who do not ovulate by day 28 receive oral clomiphene citrate daily on days 36-40.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Obese women with chronic anovulation due to polycystic ovary syndrome (PCOS)

Must have oligoamenorrhea and hyperandrogenemia

--Prior/Concurrent Therapy--

At least 2 months since prior standard therapy (including over the counter drugs) At least 2 months since prior investigational agents

--Patient Characteristics--

Hematopoietic: Hematocrit greater than 38%

Hepatic: Liver function normal No clinically significant hepatic disease

Renal: No clinically significant renal disease Creatinine less than 1.4 mg/dL No proteinuria

Cardiovascular: No clinically significant cardiac disease

Pulmonary: No clinically significant pulmonary disease

Hormonal: Thyroid function normal Prolactin normal Fasting 17 alpha-hydroxy progesterone less than 200 mg/dL OR No late onset adrenal hyperplasia 21 alpha-hydroxylase deficiency

Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception No diabetes mellitus No clinically significant neurologic, psychiatric, infectious, neoplastic, or metabolic disease No clinically significant malignant disease except nonmelanomatous skin cancer At least 1 year since any prior drug abuse or alcoholism

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: William S. Evans, Study Chair — University of Virginia